CLINICAL TRIAL: NCT04639167
Title: Volunteer-led "Paths to Everyday Life" (PEER) Peer Support Group Intervention to Adults With Mental Health Difficulties Versus Service as Usual in the Community - Results From a Randomized Two-armed, Multi-municipal, Superiority Trial
Brief Title: Paths to Everyday Life (PEER) - a Community-based Peer Support Intervention
Acronym: PEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Collaborators: The Peer partnership association (Unknown)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEER
Record Dates: First submitted 2020-11-13; First posted 2020-11-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Impairment; Peer Group; Mental Health Disorder; Problems Psychosocial
Keywords: Peer support; Community-based; Randomized Controlled Trial; Individual companionship; Volunteer peers; Peer group sessions
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: A randomized, two-arm, investigator initiated, multi municipal, parallel-group superiority trial comparing the effect on self-reported personal recovery of the following interventions: (1) 10-week group-based peer support intervention "Paths to everyday life" (PEER) added to servide as usual (SAU) and (2) SAU alone
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants, the local coordinators and the volunteer peers cannot be blinded to the group allocation. The REDCap randomization tool will be used to facilitate randomization. To ensure concealment, the randomization schedule is stored away from the research team and the block sizes are not disclosed. The allocation is performed by a not-blinded research coordinator, who informs the participants allocated to the control group through a central telephone. Moreover, the research coordinator informs the local coordinators in each municipality about participants allocated to the intervention group through submitting the record id via secure email. The local coordinators will be able to identify the participants through their access to REDCap. The researchers will be blinded to group allocation during the process of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paths to everyday life (PEER) (Experimental): The Paths to everyday life (PEER) intervention added to service as usual (SAU) consists of a 10-week group course and an opportunity of individual companionship to persons with mental vulnerability and mental health difficulties. The 10 week group sessions is facilitated by two volunteer peers with their own lived experiences with mental vulnerability.
  Interventions: Behavioral: Paths to everyday life (PEER)
- Service as usual (SAU) (No Intervention): Participants who will be allocated to the control group of the trial will receive service as usual (SAU) by their social security officer, or no specific service if the participant has been referred to the trial by self-referral. Participants who are referred to the trial via §82 in the municipality, can receive other §82 offers depending on the individual municipality.

INTERVENTIONS:
Behavioral: Paths to everyday life (PEER) — The intervention consists of a 10-week group course and the opportunity of individual companionship to e.g. local activities in civil society, municipal social services, education, health and employment. The 10-week group sessions are delivered by two volunteer peers with their own experiential knowledge of mental vulnerability and mental health difficulties. The aim is to form a constructive community through group sessions where exchanges of lived experiences, mutuality and opportunities for social network development can develop.
  Arms: Paths to everyday life (PEER)

SUMMARY:
The aim of this randomized, two-arm, investigator initiated, multi municipal, parallel-group superiority trial is to compare the effect on self-reported personal recovery of the following interventions: (1) 10-week group-based peer support intervention "Paths to everyday life" (PEER) added to service as usual (SAU); and (2) SAU alone. The primary outcome is self-reported personal recovery at end of intervention. Secondary and exploratory measures include empowerment, quality of life, functioning, hope, self-efficacy, self-advocacy and social network. The investigators, hypothesize that the superiority of the PEER intervention will be applicable for secondary outcomes and exploratory measures at end of intervention so that improvement in empowerment, hope, self-efficacy, self-advocacy, social network, quality of life and functioning will be improved among participants allocated to the PEER intervention.

DETAILED DESCRIPTION:
The "Paths to everyday life" (PEER) intervention is a newly developed community-based peer support intervention targeting persons with mental vulnerability and mental health difficulties. The development of the PEER intervention is conducted in a collaboration between the Peer partnership association and the Copenhagen Research Center for Mental Health (CORE), Recovery & Inclusion, Mental Health Center Copenhagen.

The PEER intervention is inspired from: Peer support groups in the MIND Leeds organization; Manuals for peer support services and peer training, which has shown positive effect on measures of personal recovery in RCTs; Practical guides to everyday life developed by consumers of mental health treatment in Denmark; and lived experiences of mental illness and recovery within the project group. The content of the ten group sessions is developed from themes identified in the CHIME (Connectedness; Hope; Identity; Meaning; Empowerment) framework as promoting the personal recovery process, as well as knowledge from systematic reviews and meta-analyses in the field focusing on the effect of peer support. The entire PEER intervention is described in a comprehensive manual and detailed instructions have been prepared for the volunteer peers to make it accessible and ensure similarity across the groups. The manual of the PEER intervention has been further developed in a pilot study of the 10 week group sessions in a qualitative evaluation (N=25) in the period Feb.-Sept. 2020 in the collaborative municipalities Copenhagen, Elsinore and Fredericia.

The PEER intervention consists of a 10-week group course and the opportunity of individual companionship to e.g. local activities in civil society, municipal social services, education, health and employment. It is mandatory for the participants to participate in an introductory meeting with the purpose of informing about the group process, the individual companionship and the RCT, so that participation in the intervention becomes the participants' own informed choice. The group sessions are delivered by two volunteer peers with their own experiental knowledge of mental vulnerability and personal recovery. The volunteer peers must complete a basic peer education to facilitate the group course and enter individual companionship. A fidelity scale is developed and used for biannual fidelity reviews to ensure intervention program adherence and continuous focus on program implementation and improvement.

The overall purpose of the PEER intervention is to find a way to live life in a meaningful, energizing way - despite still finding some things challenging. The aim is to form a constructive community through group sessions where exchanges of lived experiences, mutuality and opportunities for social network development can form. The investigators hypothesize, that the volunteer peers by sharing their own experiences with mental vulnerability and personal recovery can create trust and inspire the participants to safely share their own experiences. Additionally, that the volunteer peers by presenting group themes and by participating on an equal footing with the participants in the group exercises can contribute to the participants' experience of connectedness with others, as well as promote the participants self-esteem and belief in possibilities, dreams and aspirations to regain meaning in life circumstances, control and responsibility for own life.

The PEER intervention will be evaluated in a two armed randomized controlled trial. The primary hypothesis for the trial is that participants allocated to the PEER intervention added to service as usual (SAU) gain a significantly increased experience of self-reported personal recovery at end of intervention than participants who are allocated to SAU alone.

The PEER intervention is not expected to have any severe side effects. However, when trial recruitment and the intervention phase has ended, safety measures i.e. number of somatic and psychiatric hospitalization days, death, suicide and probable self-harm is obtained from the Danish central registers to examine any severe adverse effects during the intervention period.

The sample size and power calculations was conducted using PS Power and Sample Size Calculations software. With an allocation ratio of 1:1 and a minimum clinically relevant difference of 5, a power of 80% and a significance level of 0.05%, we need 284 participants, i.e. 142 in the intervention group and 142 in the control group in order to reject the null hypothesis that self-assessed personal recovery is equal in the control group and the PEER group. Data analyzes will be based on the intention-to-treat principle i.e. that data from all participants will be included corresponding to the group to which the participants have been allocated. In case of missing data, multiple multivariate imputations will be used.

ELIGIBILITY:
Inclusion Criteria:

* Citizens using the municipal social service in the participating municipalities for support and assistance due to mental vulnerability and mental health difficulties, corresponding to the target group for §82 in the law of social service - i.e. citizens diagnosed with a mental illness and/or who is affected by mental dissatisfaction to a degree that limits the unfolding of life. Additionally, citizens who self-refer to the trial with similar mental health challenges.
* Are residents of collaborating municipalities at baseline.
* Can understand, speak, and read Danish.
* Are aged 18 years or older.
* Have given verbal and written consent to participate in the trial.

Exclusion criteria:

1. Citizens intoxicated by alcohol and/or other substances - if they according to the local coordinator's judgment cannot participate in the peer group, they are advised to contact professional help.
2. Citizens with specific suicide plans - if they according to the local coordinator's judgment cannot participate in the peer group, they are advised to contact professional help.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Questionnaire about the Process of Recovery (QPR-15) | At end of intervention (3 months)
  Personal recovery is measured with the Questionnaire about Process of Recovery (QPR-15), which consist of 15 items measuring aspects of personal recovery i.e. experiences of connectedness, hope, identity, meaning and empowerment - based on mental health consumer experiences of recovery. In psychometric evaluations, QPR-15 demonstrated good internal consistency and test-retest reliability, as well sufficient convergent validity and moderate sensitivity to change. Each item is scored on a 5-point Likert scale ranging from 0 (strongly disagree) to 5 (strongly agree) and gives a total score between 0-60.

SECONDARY OUTCOMES:
The Empowerment Scale, Rogers (ESR) | At end of intervention (3 months)
  Empowerment is measured with The Empowerment scale Rogers (ESR), which consist of 28 items measuring a person's resources, opportunities and sense of control over their own life - based on mental health consumer experiences of empowerment. The Empowerment scale is widely used and validated and is scored on a 4-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree)
The Manchester Short Assessment of Quality of life (MANSA) | At end of intervention (3 months)
  Quality of life is measured with The Manchester Short Assessment of Quality of life (MANSA), which consist of 16 items whereas 4 items measure objective quality of life (close relationships, contact with friends, crime and assault) and 12 items measure subjective quality of life (satisfaction with life as a whole, work, financial situation, friendships, leisure activities, housing, personal safety/security, cohabitation, sex life, family relationships and health). The questionnaire has been validated and is scored on a 7-point scale ranging from 1 (couldn't be worse) to 7 (couldn't be better).
Work and Social Adjusment Scale (WSAS), | At end of intervention (3 months)
  Functioning is measured with the Work and Social Adjusment Scale (WSAS), which is a 5-item self-reported questionnaire covering a person's perceived functioning in terms of the domains 1) Workability; 2) Performing tasks at home (cleaning, shopping, paying bills, etc.); 3) Social leisure activities (parties, dating, tours, visits, cinema, etc.); 4) private leisure activities (reading, gardening, sewing, walking alone, etc.) and; 5) Ability to form and maintain close relationships. The questionnaire is widely used and validated and scored on an 8-point scale ranging from 0 (not at all) to 8 (very seriously).

OTHER OUTCOMES:
General Self-efficacy (GSE) | At end of intervention (3 months)
  Self-efficacy is measured with the general self-efficacy scale (GSE), which consists of 10-items designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. The GSE scale is widely used and validated and is scored on a 4-point Likert scale ranging from 0 (not at all true) to 4 (exactly true).
The Self-advocacy scale (SAS) | At end of intervention (3 months)
  Self-advocacy is measured with the self-advocacy scale (SAS), which consists of 8-items involving taking care of yourself, being organized and prepared, finding the resources you need, and communicating and negotiating to get your needs met. The SAS scale is only used and validated in research about acquired brain injury and scored on a 4-point Likert scale ranging from 0 (not confident) to 4 (very confident).
State Hope Scale (SHS) | At end of intervention (3 months)
  Hope is measured with the State Hope Scale (SHS), which consist of 6-items measuring hope ie the belief in one's own ability to initiate and maintain actions and ways to achieve goals. The state hope scale is widely used and validated and scored on an 8-point scale ranging from 1 (definitely false) to 8 (definitely true).
Copenhagen Social Relations Questionnaire (CSRQ) | At end of intervention (3 months)
  Social network is measured with a modified version of the Copenhagen Social Relations Questionnaire (CSRQ), which consist of 19-items covering frequency of social contact, social support in everyday life, quality of social relations and frequency of participating in local social activities. The questionnaire has satisfactory validity and reliability and is widely used in Danish population surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, MD PhD, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data that support the findings in this article will be made available after de-identification, along with the statistical analysis plan, upon reasonable request from researchers who provide a methodologically sound proposal. To request access, proposals should be directed to the corresponding author. Data requestors will need to sign a data access agreement to gain access to the data. The register-based data cannot be provided on request because it is hosted by Statistics Denmark. The data was only accessible to researchers connected to the project, and it was not possible to download the final trial data set.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available in 5 years from publication of the results.
Access Criteria: To request access, proposals should be directed to the corresponding author. Data requestors will need to sign a data access agreement to gain access to the data.

REFERENCES:
- [Background] Pitt V, Lowe D, Hill S, Prictor M, Hetrick SE, Ryan R, Berends L. Consumer-providers of care for adult clients of statutory mental health services. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD004807. doi: 10.1002/14651858.CD004807.pub2. PMID 23543537
- [Background] Fuhr DC, Salisbury TT, De Silva MJ, Atif N, van Ginneken N, Rahman A, Patel V. Effectiveness of peer-delivered interventions for severe mental illness and depression on clinical and psychosocial outcomes: a systematic review and meta-analysis. Soc Psychiatry Psychiatr Epidemiol. 2014 Nov;49(11):1691-702. doi: 10.1007/s00127-014-0857-5. Epub 2014 Mar 17. PMID 24632847
- [Background] Lloyd-Evans B, Mayo-Wilson E, Harrison B, Istead H, Brown E, Pilling S, Johnson S, Kendall T. A systematic review and meta-analysis of randomised controlled trials of peer support for people with severe mental illness. BMC Psychiatry. 2014 Feb 14;14:39. doi: 10.1186/1471-244X-14-39. PMID 24528545
- [Background] Gillard S, Gibson SL, Holley J, Lucock M. Developing a change model for peer worker interventions in mental health services: a qualitative research study. Epidemiol Psychiatr Sci. 2015 Oct;24(5):435-45. doi: 10.1017/S2045796014000407. Epub 2014 Jul 3. PMID 24992284
- [Background] Repper J, Carter T. A review of the literature on peer support in mental health services. J Ment Health. 2011 Aug;20(4):392-411. doi: 10.3109/09638237.2011.583947. PMID 21770786
- [Background] Walker G, Bryant W. Peer support in adult mental health services: a metasynthesis of qualitative findings. Psychiatr Rehabil J. 2013 Mar;36(1):28-34. doi: 10.1037/h0094744. PMID 23477647
- [Background] Williams J, Leamy M, Pesola F, Bird V, Le Boutillier C, Slade M. Psychometric evaluation of the Questionnaire about the Process of Recovery (QPR). Br J Psychiatry. 2015 Dec;207(6):551-5. doi: 10.1192/bjp.bp.114.161695. Epub 2015 Oct 8. PMID 26450585
- [Background] Chien WT, Clifton AV, Zhao S, Lui S. Peer support for people with schizophrenia or other serious mental illness. Cochrane Database Syst Rev. 2019 Apr 4;4(4):CD010880. doi: 10.1002/14651858.CD010880.pub2. PMID 30946482
- [Background] Leamy M, Bird V, Le Boutillier C, Williams J, Slade M. Conceptual framework for personal recovery in mental health: systematic review and narrative synthesis. Br J Psychiatry. 2011 Dec;199(6):445-52. doi: 10.1192/bjp.bp.110.083733. PMID 22130746
- [Background] Law H, Neil ST, Dunn G, Morrison AP. Psychometric properties of the questionnaire about the process of recovery (QPR). Schizophr Res. 2014 Jul;156(2-3):184-9. doi: 10.1016/j.schres.2014.04.011. Epub 2014 May 9. PMID 24816049
- [Background] Rogers ES, Chamberlin J, Ellison ML, Crean T. A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatr Serv. 1997 Aug;48(8):1042-7. doi: 10.1176/ps.48.8.1042. PMID 9255837
- [Background] Rogers ES, Ralph RO, Salzer MS. Validating the empowerment scale with a multisite sample of consumers of mental health services. Psychiatr Serv. 2010 Sep;61(9):933-6. doi: 10.1176/ps.2010.61.9.933. PMID 20810594
- [Background] Bjorkman T, Svensson B. Quality of life in people with severe mental illness. Reliability and validity of the Manchester Short Assessment of Quality of Life (MANSA). Nord J Psychiatry. 2005;59(4):302-6. doi: 10.1080/08039480500213733. PMID 16195135
- [Background] Priebe S, Huxley P, Knight S, Evans S. Application and results of the Manchester Short Assessment of Quality of Life (MANSA). Int J Soc Psychiatry. 1999 Spring;45(1):7-12. doi: 10.1177/002076409904500102. PMID 10443245
- [Background] Thandi G, Fear NT, Chalder T. A comparison of the Work and Social Adjustment Scale (WSAS) across different patient populations using Rasch analysis and exploratory factor analysis. J Psychosom Res. 2017 Jan;92:45-48. doi: 10.1016/j.jpsychores.2016.11.009. Epub 2016 Nov 30. PMID 27998511
- [Background] Luszczynska A, Scholz U, Schwarzer R. The general self-efficacy scale: multicultural validation studies. J Psychol. 2005 Sep;139(5):439-57. doi: 10.3200/JRLP.139.5.439-457. PMID 16285214
- [Background] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Background] Hawley L, Gerber D, Pretz C, Morey C, Whiteneck G. Initial validation of personal self-advocacy measures for individuals with acquired brain injury. Rehabil Psychol. 2016 Aug;61(3):308-316. doi: 10.1037/rep0000093. Epub 2016 May 12. PMID 27177213
- [Background] Lund R, Nielsen LS, Henriksen PW, Schmidt L, Avlund K, Christensen U. Content validity and reliability of the Copenhagen social relations questionnaire. J Aging Health. 2014 Feb;26(1):128-50. doi: 10.1177/0898264313510033. PMID 24584264
- [Background] Deegan PE. The lived experience of using psychiatric medication in the recovery process and a shared decision-making program to support it. Psychiatr Rehabil J. 2007 Summer;31(1):62-9. doi: 10.2975/31.1.2007.62.69. PMID 17694717
- [Background] Anthony WA. Recovery from mental illness: The guiding vision of the mental health service system in the 1990s. Psychosoc Rehabil J. 1993;16(4):11-23.
- [Background] Poulsen CH, Egmose CH, Ebersbach BK, Hjorthoj C, Eplov LF. A community-based peer-support group intervention "Paths to EvERyday life" (PEER) added to service as usual for adults with vulnerability to mental health difficulties - a study protocol for a randomized controlled trial. Trials. 2022 Sep 2;23(1):727. doi: 10.1186/s13063-022-06670-6. PMID 36056407
- [Derived] Poulsen CH, Egmose CH, Ebersbach B, Hjorthoj C, Eplov LF. The "Paths to everyday life" peer support intervention for adults with mental health difficulties versus service as usual in a Danish community setting - results from a randomized two-armed, multi-site, superiority trial. BMC Psychiatry. 2025 Jul 11;25(1):695. doi: 10.1186/s12888-025-07011-y. PMID 40646520
- [Derived] Poulsen CH, Egmose CH, Bjorkedal SB, Eplov LF. Intervention delivery in the 'Paths to everyday life' (PEER) trial: a qualitative study of the perspectives of the peer volunteers with lived experiences of being in personal recovery of mental health difficulties. BMC Psychiatry. 2025 Jul 2;25(1):671. doi: 10.1186/s12888-025-06982-2. PMID 40604516
- [Derived] Egmose CH, Poulsen CH, Bjorkedal SB, Eplov LF. The 'Paths to everyday life' (PEER) trial - a qualitative study of mechanisms of change from the perspectives of individuals with mental health difficulties participating in peer support groups led by volunteer peers. BMC Psychiatry. 2024 Aug 13;24(1):555. doi: 10.1186/s12888-024-05992-w. PMID 39138435

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT04639167/SAP_001.pdf